CLINICAL TRIAL: NCT00530400
Title: Prospective, Double-Blind, Randomized, Placebo-Controlled Trial of Single-Dose Cefuroxime Prophylaxis in Herniated Disk Surgery
Brief Title: Study of the Efficacy of Preoperative Cefuroxime Prophylaxis to Prevent Surgical Site Infection in Herniated Disk Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University Hospital, Geneva (Other); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CFX93LS06
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Surgical Wound Infection
Keywords: Antibiotic prophylaxis; Bacterial Infections / prevention & control; Surgical wound infection / prevention & control; Neurosurgery; Postoperative Complications / prevention & control; Clinical trial [publication type]
MeSH Terms: conditions — Surgical Wound Infection; Bacterial Infections; Postoperative Complications | interventions — Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): intravenous 1.5g cefuroxime
  Interventions: Drug: cefuroxime
- 2 (Placebo Comparator): intravenous placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cefuroxime — preoperative intravenous 1.5g cefuroxime
  Arms: 1
Drug: placebo — preoperative intravenous placebo
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether a single, pre-operative dose of cefuroxime is effective in preventing surgical site infection in patients undergoing surgery for herniated disk

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18
* spinal surgery for herniated disk

Exclusion Criteria:

* known or suspected hypersensitivity to cephalosporins
* type I hypersensitivity to betalactamic antibiotics
* severe renal function impairment
* acquired immune deficiency syndrome (AIDS) or other conditions of severe immuno-suppression
* antibiotic therapy for concomitant infection at the time of surgery
* pregnancy
* refusal to participate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1369 (Actual)
Dates: Start 1994-04; Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of a surgical site infection | 6 months

SECONDARY OUTCOMES:
Occurrence of a post-operative infection other than surgical site infection | 6 monts
Serious adverse event | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Francioli, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Switzerland (2):
  - Hôpitaux Universitaire de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne